CLINICAL TRIAL: NCT04199195
Title: A Longitudinal Study in a Cohort Aged 60 Years and Older to Obtain Mechanistic Knowledge of the Role of the Gut Microbiome During Normal Healthy Ageing in Order to Develop Strategies That Will Improve Lifelong Health and Wellbeing.
Brief Title: Microbiome of the Ageing Gut and Its Effect on Human Gut Health and Cognition.
Acronym: MOTION
Status: Active, not recruiting | Type: Observational
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: QIB04-2018
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Ageing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool, blood and colon tissue biopsies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Males and females aged at least 60 years.: A longitudinal study of one cohort of 360 participants aged at least 60 years. Participants will be required to provide a stool sample, provide a blood sample and complete a health questionnaire every 6 months for 4 years. At alternate visits, participants will be required to under go cognitive assessments and physical measurements.
  Participants will be required to under go an Optical Coherence Tomography Scan 3 times over 4 years.
  Sub group 1 - During a routine care colonoscopy, at least 90 participants will have 6-8 colon tissue biopsies taken for research purposes.
  Sub group 2 - Participants from cohort 3 only will be offered an optional brain MRI until the required number of 30 participants is achieved.

SUMMARY:
The investigators aim to undertake a 49-month longitudinal study in a cohort of 360 healthy individuals of 60 years and older, living in East Anglia to understand the role of gut microbes (the microbiome) in healthy ageing. The investigators also aim to identify changes in the structure and function of the gut microbe populations that are associated with deteriorating mental health and cognitive function. Using clinically validated cognitive assessments and tests, study participants will be stratified in to one of three risk groups for developing dementia:-

Cohort 1 - low (n=120). Cohort 2 - medium (n=120). Cohort 3 - high (n=120).

Participants will be recruited from three streams - Primary Care, The NHS Bowel Cancer Screening Programme (BCSP) and the Norfolk & Suffolk Foundation Trust (NSFT).

Following initial Telephone Contact and the Pre-Study Visit, all participants will be required to attend the Quadram Institute Clinical Research Facility (QI CRF) every 6 months over 4 years. At each of these follow-up visits, the participant will provide a stool sample (collected at home) and at differing time points, provide a blood sample and undergo a series of physical measurements, cognitive tests/questionnaires and complete a health questionnaire. All participants will undergo Optical Coherence Tomography scans at the Beccles & District War Memorial Hospital.

There will be 2 subgroups in this study.

Subgroup 1 - at least 30 participants from each cohort (n= at least 90) will undergo colonic tissue biopsies as part of routine clinical care using the NHS BCSP.

Subgroup 2 - 30 participants from Cohort 3 will undergo brain imaging at the Norfolk & Norwich University Hospital (NNUH) Imaging Department.

The results of the study will provide new insights into the gut-brain axis and the relationship between age-associated changes in gut microbe populations and declining mental health. Such insights will be of enormous value in developing new microbe-based strategies to improve lifelong health and wellbeing that impact on dementia development.

DETAILED DESCRIPTION:
Humans have co-evolved with populations of colonising microbes and their genomes to establish a mutually beneficial relationship. The gut microbiome represents the largest population of resident microbes in humans and is highly diverse and plays essential roles in digestion and pathogen protection. Perturbations in populations of gut bacteria (dysbiosis or dysbacteriosis) in response to, for example, infections or drugs, have been associated with an increased risk of various chronic diseases including obesity, cancer and inflammatory bowel disease (IBD).

In older individuals an array of complex and characteristic clinical changes that includes a basal proinflammatory state (so called "inflammaging"), can directly interface with gut microbes of older adults that can enhance susceptibility to diseases accompanying aging, and reduce healthy lifespan. Studies in older adults demonstrate that the makeup and functional attributes of the intestinal microbiota correlates with lifestyle (e.g. diet and location of residence) and behaviour (e.g. medications), and basal level of inflammation. Links exist between the intestinal microbiota and a variety of clinical problems plaguing older adults, including physical frailty, Clostridium difficile colitis, vulvovaginal atrophy, colorectal carcinoma, and atherosclerotic disease. These links are however, principally associative with very little evidence of causality.

The gut microbiome establishes a mutualistic relationship with its host and contributes to maintaining homeostasis. Its composition can be influenced and changed by numerous host (e.g. genome, age), environmental (e.g. diet, medicines, infections), and lifestyle and behavioural factors (e.g. travel, habitat). Changes in the structure and/or function of the microbiome (dysbiosis) can result in damage to, or infection of, barrier epithelial cells enabling microbes and microbial products to cross the compromised barrier and gain access to underlying tissues and immune cells, leading to immune activation and (chronic) inflammation.

Age is a major risk factor for the development of cognitive dysfunction with dementia being one of the most common disorders linked to ageing. Dementia affects an estimated 47 million people worldwide and is projected to affect over 131 million people by 2050. Cognitive function declines with age, ranging from relatively minor everyday slips of action, through subjective cognitive decline, mild cognitive impairment (MCI), then to major or mild neurocognitive disorder/dementia in some instances. Up to 50% of those with MCI are predicted to develop dementia within 5 years.

The development of new treatments to prevent dementia is hindered by a lack of predictive biomarkers. The gut microbiome is a potential marker for progressive declining intrinsic capacity, which is a composite of all the physical and mental attributes on which an individual can draw, not only in older age but across their lives. Evidence of age-associated changes in the gut microbiome comes from population-based studies, one of the largest and most comprehensive was ELDERMET, a study that examined the faecal microbiome of elderly individuals living in the community or in care homes in Ireland. The results identified differences in the composition of the gut microbiome of elderly individuals compared with younger individuals, and that these differences were associated with poorer health status in the elderly (e.g. poor dentition, dysphagia, loss of salivation, decreased physical activity and constipation).

However, in relying on data from samples taken at a single timepoint, this study provides only a 'snapshot' of what is happening but little insight into the dynamics or stability of any changes in the gut microbiome over time in different individuals or groups of participants. It is also impossible to determine whether the changes noted are drivers or consequences of unhealthy ageing. In addition, this study did not include assessments of mental health and cognitive function, which are major comorbidities associated with ageing. The fact that structural changes within the gut microbiome occur during ageing is a consistent finding across different studies. However, the scale and nature of the changes noted vary considerably between studies, and amongst individuals within the same study. Larger longitudinal studies with sequential (serial) sampling of the gut microbiome during ageing would provide a clearer picture of how the gut microbiome changes during ageing, and whether it is a contributing factor to declining health in old age and/or in the development of neurodegenerative disorders and dementia.

The link between potentially pathogenic changes in the gut microbiome (dysbiosis) in individuals with neurodegenerative disorders comes mainly from observational studies in patients with Alzheimer's (AD) or Parkinson's disease (PD), and from animal (rodent) models. Analysis of the faecal microbiome of dementia patients has identified an increased prevalence of Prevotellaceae and Enterobacteriaceae species in PD, and an increased prevalence of Clostridia, Bacteroides and Verrucomicrobia species in AD patients. compared with healthy individuals. In addition, many PD and AD patients reported gut symptoms including irritable bowel syndrome prior to neurological symptoms developing. Furthermore, antibiotic treatment to eradicate gut pathogens (e.g. H. pylori) can improve L-dopa action and reduce clinical symptoms in PD patients. Perhaps the most compelling evidence for a causal link between gut microbes and neurodegenerative disease comes from the finding that, when faecal microbiomes from PD patients are transferred into PD-susceptible mice, symptom development accelerates and the mice suffer greater motor dysfunction than control mice receiving faecal microbiomes of healthy individuals. Although collectively these findings implicate the gut microbiome in the pathogenesis of neurodegenerative disorders, the studies carried out to date have failed to identify which species of bacteria (or any other member of the gut microbiome; viruses, archaea, fungi, protozoa) are critically important for mental health and in the development of dementia, when during ageing do changes in the population size and/or function of critical species occur, and once established how do these critical species influence brain signalling, neuroinflammation and pathology?

Subgroup 1 - Colon tissue biopsy (n= at least 90). Microbe populations that are specifically and intimately associated with the lining of the gut wall are ideally situated to influence the host and intestinal cells, but they can be underrepresented or absent in stool samples. For this reason, colon tissue samples are important to: 1) fully identify the microbes that are in most intimate contact with the host 2) identify and analyse how the cells within the tissue respond and react to these microbes and their products.

6-8 pinch biopsies each measuring 3mm cubed will be taken for research biopsies from the large bowel during the routine care colonoscopy (these will taken in addition to routine care biopsies). The research biopsies are taken to examine the microbiome that is adhering directly to the mucosal lining of the colon.

Subgroup 2 - Brain MRI scans (n=30 from cohort 3). Scans will be performed to allow for the cognitive and behavioural data collected at the previous visits to be related to neuroanatomical changes. The 60-minute scan will capture both structural and functional sequences. Structural sequences will allow measurement of grey and white matter integrity in participants, whereas functional sequences will allow measurement of brain connectivity and perfusion changes. We hypothesize that medial temporal structures will be intact in low risk participants but those in the medium risk group might already show subtle structural and functional changes.

Another screening test with potential as a biomarker for ageing and dementia development is retinal morphometry. The retina is the only part of the central retinal nervous system that can be directly visualized. Optical Coherence Tomography (OCT) is a rapid, non-invasive imaging tool that can produce 3- dimensional cross-sectional images of the retina, and permits precise and accurate measurement of the thickness of individual retinal components. The retinal nerve fiber layer (RNFL) is the innermost layer of the retina and is comprised of the retinal ganglion cell axons, which link the outer neuroretina to the dorsal lateral geniculate nucleus, where synaptic connections lead to the visual cortex. In a very recent multi-centre study of individuals aged between 40 and 69 years of age, OCT imaging revealed that a thinner RNFL was associated with worse cognitive function in individuals with no neurodegenerative disease; it was also associated with a greater likelihood of subsequent cognitive decline. This makes a strong case for regarding retinal anatomical measures as a potentially useful screening marker to identify those at risk of developing dementia.

The studies carried out to date highlight the need to develop a more holistic and integrated understanding of human ageing: There is a need to understand how (or whether) changes in one organ system (e.g. the gut) are related to changes occurring elsewhere in the body (e.g. in the brain). In order to begin to answer these fundamentally important questions, the investigators have designed the MOTION study to obtain a clearer picture of how the gut microbiome changes during ageing in a cohort over the age of 60 years without existing serious medical conditions at the point of study consent, and how these changes relate to declining intrinsic capacity and increasing cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged at least 60 years.
* Must be able to provide informed consent.
* Must be able to complete the Cognitive Tests/Questionnaires, Health Questionnaires by themselves and be familiar with using an ipad/tablet.

Exclusion Criteria:

* Currently taking part in an interventional study.
* Living with or related to any member of the research team.
* Have a diagnosis of Dementia, Parkinson's Disease, Alzheimer's Disease, Creutzfeldt-Jakob disease (CJD), Picks Disease.
* Bipolar Disorder.
* Obsessive Compulsive Disorder.
* Untreated current clinical depression.
* Have irreversible brain injury.
* Have had a stroke.
* Have epilepsy.
* Take more than a daily dose of probiotics.
* Have a long-standing gastrointestinal or liver function abnormality requiring on- going medical management or medication.
* History of cancer within the last 5 years except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision.
* Unstable dietary history as defined by major changes in diet during the previous month, where a major food group in the diet has been stopped or significantly increased, for example become vegetarian, vegan or stopped eating red meat.
* History of alcohol, drug or substance abuse. History of Hepatitis B or Hepatitis C.
* Major surgery of the gastrointestinal tract, apart from gall bladder or appendix removal, in the past five years.
* Any major bowel resection at any time.
* History of Ulcerative Colitis, Crohn's Disease or Diverticulitis.
* Persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhoea of unknown cause, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated).
* Constipation.
* Regular use of laxatives.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females aged at least 60 years without existing serious health conditions at the point of providing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Microbial composition | 48 months
  Changes in microbiome measured by DNA/RNA sequencing of longitudinal samples collected at 6 monthly intervals.

SECONDARY OUTCOMES:
Establishment of a biorepository | 48 months
  Banking of longitudinal samples collected throughout the study that will be used in future research.
Microbial signatures identified and correlated with measures of declining health and (organ) functionality. | 48 months
  Changes in microbial composition associated with cognitive function and clinical data collected throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Simon R Carding, PhD, Study Chair — Quadram Institute Bioscience; Simon M Rushbrook, MBBS, Principal Investigator — Norfolk & Norwich University Hospital; Michael Hornberger, PhD, Principal Investigator — University of East Anglia; Janak Saada, MBBS, Principal Investigator — Norfolk & Norwich University Hospital; Ben Burton, FRC Opth, Principal Investigator — James Paget Hospital
Locations (1):
- Quadram Institute Bioscience, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study team will ensure fully compliance with the standards required for deposition of information in any relevant public databases. Anonymised datasets will be kept indefinitely and available to other researchers to comply with journal requirements when required.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available at the end of the study
Access Criteria: Chief Investigator will review requests.

REFERENCES:
- [Derived] Phillips S, Watt R, Atkinson T, Rajan S, Hayhoe A, Savva GM, Hornberger M, Burton BJL, Saada J, Cambell-Kelly M, Rushbrook S, Carding SR. A protocol paper for the MOTION Study-A longitudinal study in a cohort aged 60 years and older to obtain mechanistic knowledge of the role of the gut microbiome during normal healthy ageing in order to develop strategies that will improve lifelong health and wellbeing. PLoS One. 2022 Nov 18;17(11):e0276118. doi: 10.1371/journal.pone.0276118. eCollection 2022. PMID 36399457